CLINICAL TRIAL: NCT07336459
Title: AI-Driven Multimodal Rehabilitation Framework for Type 2 Diabetes Integrating Digital Health Technologies, Intermittent Fasting, and Resistance Training to Optimize Metabolic and Functional Outcomes
Brief Title: AI-Driven MRF Type 2 Diabetes Integrating DHT IF and Resistance Training to OM and Functional Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PhDRSW/Batch-Fall23/2228
Record Dates: First submitted 2025-11-21; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus 1
MeSH Terms: conditions — Diabetes Mellitus, Noninsulin-Dependent, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Guided Multimodal Rehabilitation Program (Experimental)
  Interventions: Combination Product: AI-Guided Multimodal Rehabilitation Program
- Standard Diabetes Care (Active Comparator)
  Interventions: Diagnostic Test: Standard Diabetes Care

INTERVENTIONS:
Combination Product: AI-Guided Multimodal Rehabilitation Program — Digital Health: Mobile AI-based app with glucose tracking, exercise reminders, and fasting compliance monitoring Intermittent Fasting: 16:8 time-restricted feeding protocol, 5 days/week Resistance Training: 3 sessions/week (45 minutes), supervised + home-based program using elastic bands & bodyweight
  Arms: AI-Guided Multimodal Rehabilitation Program
Diagnostic Test: Standard Diabetes Care — Usual pharmacological treatment + general lifestyle advice No structured AI, fasting, or exercise protocol
  Arms: Standard Diabetes Care

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of an AI-driven multimodal rehabilitation framework combining digital health technologies, intermittent fasting, and resistance training in individuals with Type 2 Diabetes Mellitus (T2DM). The study will integrate mobile-based AI monitoring for glucose trends, physical activity tracking, and dietary adherence reminders, thereby improving patient engagement and self-management.

DETAILED DESCRIPTION:
Participants will be randomized into two groups: the intervention group receiving AI-guided resistance training alongside intermittent fasting, and the control group receiving standard diabetes care. Outcomes will include changes in HbA1c, insulin sensitivity (HOMA-IR), muscle strength, functional mobility, and quality of life. The study will also assess adherence, feasibility, and cost-effectiveness. By utilizing AI-enabled technology and lifestyle-based interventions, this study addresses the gap between clinical management and sustainable self-care in T2DM. The framework is designed to be low-cost, scalable, and adaptable, making it suitable for resource-limited healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes (≥1 year)
* HbA1c between 6.5% and 9.0%
* Sedentary or low physical activity levels
* BMI: 25-35 kg/m²
* Able to perform mild-to-moderate exercise

Exclusion Criteria:

* any other disability
* not willing

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c (Biochemical Outcome) | 24 Months
  HbA1c will be assessed from venous blood and reported as a percentage (%).
HOMA-IR (Biochemical Outcome) | 24 Months
  HOMA-IR will be derived from fasting glucose and fasting insulin measurements and presented as a unitless index.
6-Minute Walk Test (Functional capacity; distance in meters) | 24 Months
  The 6-Minute Walk Test (6MWT) measures functional capacity by recording the total distance (in meters) a person can walk in six minutes on a flat, straight course. Healthy adults typically walk between 400 and 700 meters,
WHOQOL-BREF | 24 Months
  The WHOQOL-BREF is a 26-item, self-report questionnaire developed by the World Health Organization (WHO) for measuring an individual's self-perceived quality of life. It is a widely used and cross-culturally validated abbreviated version of the original, more comprehensive WHOQOL-Score 0-100
Diabetes Self-Management Questionnaire | 24 Months
  Diabetes Self-Management Questionnaire (DSMQ), first reverse the scores for any negatively worded items so higher scores consistently indicate more effective self-care. Then, sum the scores for all items to get a raw total score. This raw score can be transformed to a scale of 0-10 by dividing the raw score by the theoretical maximum and multiplying by 10 for easier interpretation and comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No